CLINICAL TRIAL: NCT06908629
Title: Addressing Social Determinants of Health (SDOH) Among Metro Detroit Cancer Survivors: A Pilot Feasibility Study (The Resource Ready Study)
Brief Title: Addressing Social Determinants of Health Among Metro Detroit Cancer Survivors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Responsible Party: Principal Investigator, Hayley Thompson, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2024-042
Record Dates: First submitted 2025-03-27; First posted 2025-04-03 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Cancer; Cancer Survivors; Gastrointestinal Cancers; Neuroendocrine Tumors; Multiple Myeloma, Neoplasms
MeSH Terms: conditions — Neoplasms; Gastrointestinal Neoplasms; Neuroendocrine Tumors; Multiple Myeloma | interventions — Referral and Consultation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Screening Needs Assessment (Experimental)
  Interventions: Other: Implementation of social determinants of health screening and referral

INTERVENTIONS:
Other: Implementation of social determinants of health screening and referral — Participants will be referred to community-based resources in response to their answers on the screening tool.

SUMMARY:
The goal of this screening study is to determine the feasibility of completing a social needs screening tool in participants who have a past or current cancer diagnosis and reside in Metro Detroit, Michigan. Main questions to answer are:

* Can we have a completion rate of at least 80% of participants filling out the screening tool?
* Can we determine procedures for patient referrals based on social needs
* Can we implement brief interventions based on food access and digital inclusion (ensuring everyone has access to the digital technologies they need to participate in society)

DETAILED DESCRIPTION:
In part 1 of the study, Participants will be administered a social screening tool either in person or via telephone. Responses to the screening tool will be translated into diagnosis codes which identify non-medical factors that may influence a patient's health status. In part 2 of the study, participants will be referred to community-based resources based on their responses to the social needs screening tool. Follow up will be made via telephone call at 2, 4, 6 and 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* past or current cancer diagnosis
* reside in metropolitan Detroit (Wayne, Oakland, Macomb counties)
* English proficient
* Actively receiving care through one of Karmano's Cancer Institute's outpatient clinics OR post treatment survivors in the Detroit Research on Cancer Survivors (ROCS) longitudinal cohort study who have reported past food insecurity and agreed to be contacted for further research

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-09-03 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants completing the screening tool | At enrollment
  80% of the 120 participants will complete the American Academy of Family Physicians (AAFP) Social Needs Screening Tool

CONTACTS AND LOCATIONS:
Locations (1):
- Karmanos Cancer Institute, Detroit, Michigan, United States